CLINICAL TRIAL: NCT00119951
Title: Health eCommunities - The Impact of Listservs on Cancer Patients
Status: Completed | Type: Observational
Sponsor: Robert Wood Johnson Foundation (Other)
Collaborators: Association of Cancer Online Resources (Other)
Other Study IDs: 49152
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Cancer
Keywords: Behavioral
MeSH Terms: conditions — Neoplasms; Behavior

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Participation on the ACOR Listserv

SUMMARY:
The purpose of this study is to assess the impact of participation in the Association of Cancer Online Resources (ACOR) mailing lists on chronic disease management for cancer patients, we are focusing on several priority areas. These include factors that influence the use of online interventions over time and the effects of patient-provider interactions on the use of eHealth interventions (as well as vice versa). We also are breaking new ground in a number of important methodological areas related to online survey research.

Our specific aims are:

1. Conduct a qualitative analysis of a 10% sample of messages (approximately 5,200) obtained over 5 months from 9 ACOR lists to develop a comprehensive set of potential chronic disease management outcomes and a fuller understanding of the issues and themes that characterize list participation. The content analysis will identify important themes and issues in the messages. These themes and issues will help in survey refinement and ground our proposed quantitative survey questionnaire items. Survey analyses will also be enriched by the qualitative data. Finally, the qualitative analysis will stand as an independent body of work.
2. Conduct a web-based survey of at least 1,680 new ACOR mailing list patient members and approximately 1,680 non-patient subscribers to assess the positive and negative effects of participation in ACOR lists at one month and four months after joining the list and completing a baseline survey.
3. Disseminate study findings to ACOR leadership, participants and the larger online community.
4. Develop a plan to convert the findings into training, recommendations, tools and policies to improve list processes. We aim to answer real world, practical questions using methodology that is at once rigorous, practical and ethical. The components are inter-related and complementary.

DETAILED DESCRIPTION:
Abstract:

Internet-based health applications can have powerful positive health effects (e.g. IOM, 2002: Eng et al., 2000; Gustafson et al., 2000). Research has focused on Internet users as consumers of information, not how they interact with one another, providing advice, consolation, encouragement and pointers to resources. There has been little evaluation of health-related mailing lists, email-based applications that connect millions of people, many with chronic diseases, with one another. The Association of Cancer Online Resources (ACOR) has teamed with The University of North Carolina (UNC) to assess the impact of participation on patients, survivors and others (including caregivers) in 15 cancer-related mailing lists managed by ACOR (www.acor.org). We are conducting a multi-method evaluation with several elements. In the qualitative component, we are conducting a content analysis of a subset of threaded discussions from archived mailing list pages to identify a comprehensive set of themes and key outcomes. This information will provide a richer understanding of mailing list processes and also will provide checks and balances on the quantitative survey. We also are evaluating the impact of being a subscriber to ACOR mailing lists on a range of outcomes by following a cohort of new subscribers for 4 months from sign-up (minimum n=1680). Baseline, one and four month web-based surveys (with telephone as an option for those who cannot do web surveys) will be administered to consenting subscribers. We also are surveying ongoing subscribers who are patients and caregivers (minimum n=1680). We will disseminate findings to several key audiences, including listowners and members as well as to a broader audience.

Project Aims:

1. Develop a comprehensive set of potential chronic disease management outcomes and a fuller understanding of the issues and themes that characterize mailing list participation.
2. Assess the effects of participation in ACOR mailing lists one month and four months after joining mailing lists and completing baseline surveys for new subscribers and through one-time surveys to ongoing subscribers and caregivers.
3. Disseminate study findings to ACOR leadership, participants and the larger online community.

Qualitative Component:

The main goal of the qualitative component is to systematically identify themes about cancer disease management and cancer mailing list support group experiences and to use that knowledge to develop a more refined understanding of mailing list use. The analyses also include:

* Participation patterns within and across mailing lists over time;
* Mailing list group processes, the nature of online group social support, and the role of mailing listowners in providing and helping group members support each other; and
* Emergent themes not previously noted in cancer-related stress and online group behavior and communication research.

Eligibility Criteria:

Eligibility is based on joining one of 15 ACOR mailing lists over a 1 ½ year accrual period. We defined eligible persons as:

* New patient/survivor subscribers aged 18 and over, have had cancer, and joined a participating mailing list within the past 10 days; or
* Ongoing patient/survivor subscribers aged 18 and over, have had cancer, and have been a member of a participating list for more than 10 days; or
* Caregiver subscribers aged 18 and over and care for a cancer patient or survivor in any capacity (actively or passively).

ELIGIBILITY:
Inclusion Criteria:

Eligibility is based on joining one of 15 ACOR mailing lists over a 1 ½ year accrual period. We defined eligible persons as:

* New patient/survivor subscribers aged 18 and over, have had cancer, and joined a participating mailing list within the past 10 days; or
* Ongoing patient/survivor subscribers aged 18 and over, have had cancer, and have been a member of a participating list for more than 10 days; or
* Caregiver subscribers aged 18 and over and care for a cancer patient or survivor in any capacity (actively or passively).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3360
Dates: Start 2003-09; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Rimer, DrPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Rimer BK, Lyons EJ, Ribisl KM, Bowling JM, Golin CE, Forlenza MJ, Meier A. How new subscribers use cancer-related online mailing lists. J Med Internet Res. 2005 Jul 1;7(3):e32. doi: 10.2196/jmir.7.3.e32. PMID 15998623
- [Result] Michael Bowling J, Rimer BK, Lyons EJ, Golin CE, Frydman G, Ribisl KM. Methodologic challenges of e-health research. Eval Program Plann. 2006 Nov;29(4):390-6. doi: 10.1016/j.evalprogplan.2006.08.011. Epub 2006 Oct 20. PMID 17950867
- [Result] Meier A, Lyons EJ, Frydman G, Forlenza M, Rimer BK. How cancer survivors provide support on cancer-related Internet mailing lists. J Med Internet Res. 2007 May 14;9(2):e12. doi: 10.2196/jmir.9.2.e12. PMID 17513283